CLINICAL TRIAL: NCT02285777
Title: A Phase 2b, Controlled, Observer-Blind, Multi-Center Study Assessing the Effectiveness, Immunogenicity and Safety of the 3rd Dose of Novartis Meningococcal ABCWY Vaccine Administered to Healthy Adolescents in the U.S.
Brief Title: Assessing the Effectiveness, Immunogenicity and Safety of Meningococcal ABCWY Vaccine Administered to Healthy Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205232; V102_16E1 (Other: Novartis Vaccines)
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-05

CONDITIONS: Meningococcal Disease
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MenABCWY Group (Experimental): Subjects who received 2 doses of MenABCWY vaccine in the parent study and a 3rd dose of MenABCWY vaccine in the current study.
  Interventions: Biological: Meningococcal ABCWY
- MenACWY Group (Active Comparator): Subjects who received 1 dose of placebo and 1 dose of MenACWY vaccine in the parent study and 1 dose of placebo in the current study.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Meningococcal ABCWY — One dose administered intramuscularly in the deltoid area of a non-dominant arm at Month 6 (Visit 1)
  Arms: MenABCWY Group
Biological: Placebo — One dose of placebo administered intramuscularly in the deltoid area of a non-dominant arm at Month 6 (Visit 1)
  Arms: MenACWY Group

SUMMARY:
This is extension of the V102_16 study (NCT02140762). V102_16E1 is designed to assess the effectiveness of a 3-dose vaccination series of MenABCWY, administered according to 0, 2, 6 month schedule, against the same panel of endemic US N. meningitidis serogroup B strains, as measured by enc-hSBA assay. The subjects who completed the parent V102_16 study will be invited at the time of their last study visit to participate in this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who completed V102_16 study and received the study vaccines as assigned in the protocol (either two doses of the MenABCWY or one dose each of MenACWY and Placebo).

Exclusion Criteria:

* Serious, acute, or chronic illnesses. Previous or suspected disease caused by N. meningitidis.
* History of any meningococcal vaccine administration other than vaccination given in the parent V102_16 protocol.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 189 (Actual)
Dates: Start 2014-12-01; Primary Completion 2015-03-26 (Actual); Study Completion 2015-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (8):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Cleveland, Ohio

REFERENCES:
- [Derived] Viviani V, Biolchi A, Pizza M. Synergistic activity of antibodies in the multicomponent 4CMenB vaccine. Expert Rev Vaccines. 2022 May;21(5):645-658. doi: 10.1080/14760584.2022.2050697. Epub 2022 Mar 14. PMID 35257644
- [Derived] Welsch JA, Senders S, Essink B, Klein T, Smolenov I, Pedotti P, Barbi S, Verma B, Toneatto D. Breadth of coverage against a panel of 110 invasive disease isolates, immunogenicity and safety for 2 and 3 doses of an investigational MenABCWY vaccine in US adolescents - Results from a randomized, controlled, observer-blind phase II study. Vaccine. 2018 Aug 23;36(35):5309-5317. doi: 10.1016/j.vaccine.2018.07.016. Epub 2018 Jul 27. PMID 30061029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 189 subjects were enrolled from 1 center in United States
Pre-assignment Details: An Interactive Response Technology (IRT) was used in the study. At Month 6 Visit of the parent study, IRT allocated the study vaccines (either MenABCWY or placebo) to the subject. Subject received either a 3rd dose of MenABCWY or one dose of a placebo, depending on their assigned vaccine group in parent study.
Period: Overall Study
Arm/Group | MenABCWY Group | MenACWY Group
Started | 95 | 94
Completed | 90 | 91
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenABCWY Group | MenACWY Group | Total
Number analyzed (Participants) | 95 | 94 | 189
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.8 (2.36) | 12.4 (2.4) | 12.6 (2.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 33 | 73
  Male | 55 | 61 | 116
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 2 | 2
  ASIAN | 1 | 0 | 1
  BLACK OR AFRICAN AMERICAN | 16 | 21 | 37
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0
  WHITE | 74 | 66 | 140
  OTHER | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects Without Bactericidal Activity at 1:4 Dilution Against Each US Neisseria Meningitides (N. Meningitidis) Serogroup B Strain at 1 Month After the 3-dose Vaccination Series.
Description: The effectiveness of three doses of MenABCWY vaccine when compared to one dose of MenACWY vaccine against a panel of US N. meningitidis serogroup B invasive disease strains at 1 month after the 3-dose vaccination series was evaluated in terms of: the combined percentage of subjects without bactericidal activity at 1:4 dilution using the human Serum Bactericidal Assay (hSBA) against each strain in MenABCWY group and MenACWY group. The data provided is an average of the percentage of subjects without bactericidal activity at 1:4 dilution across all 110 strains.
Time Frame: At Month 7 (1 month after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Effectiveness (Month 7)- included all screened subjects who provided informed consent & demographic &/or baseline screening assessments, received a subject ID & vaccination,& who provided evaluable serum sample with enc-hSBA result for at least 1 endemic N. meningitidis serogroup B invasive disease strain at Month 7.
Measure: Number; unit: Percentages of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 93 | 93
Percentages of subjects | 21.1 | 73.7
Statistical Analysis 1: Comparison: MenABCWY Group vs MenACWY Group; The Vaccine Effectiveness (VE) at 1 month after the 3-dose vaccination series for each strain is defined as [1 - (percentage of subjects without bactericidal activity at 1:4 dilution in MenABCWY group/percentage of subjects without bactericidal activity at 1:4 dilution in MenACWY group)] x 100.The combined VE across all strains was computed by mean of a generalized linear model; Test type: Other — Pre-specified; p = 0.0001, Generalized Linear Model; To obtain the VE measure which is a measure based on RR, BINOMIAL DISTRIBUTION & LOG LINK options were used to compute log10 RR & corresponding CI; Vaccine Effectiveness = 71, 95% CI 2-sided [69 to 73]

2. Secondary Outcome: Percentages of Subjects Without Bactericidal Activity at 1:4 Dilution Against Each US N. Meningitidis Serogroup B Strain at 4 Months After the 3-dose Vaccination Series.
Description: The effectiveness of three doses of MenABCWY vaccine when compared to one dose of MenACWY vaccine against a panel of US N. meningitidis serogroup B invasive disease strains at 4 months after the 3-dose vaccination series was evaluated in terms of: the combined percentage of subjects without bactericidal activity at 1:4 dilution using the hSBA against each strain in MenABCWY Group and MenACWY Group. The data provided is an average of the percentage of subjects without bactericidal activity at 1:4 dilution across all 110 strains.
Time Frame: At Month 10 (4 months after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Effectiveness (Month 10)- included all screened subjects who provided informed consent & demographic &/or baseline screening assessments, received a subject ID & vaccination, & provided evaluable serum sample with the enc-hSBA result for at least 1 endemic N. meningitidis serogroup B invasive disease strain at Month 10
Measure: Number; unit: Percentages of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 90 | 90
Percentages of subjects | 33.9 | 69.9
Statistical Analysis 1: Comparison: MenABCWY Group vs MenACWY Group; The Vaccine Effectiveness (VE) at 4 months after the 3-dose vaccination series for each strain is defined as [1 - (percentage of subjects without bactericidal activity at 1:4 dilution in MenABCWY group/percentage of subjects without bactericidal activity at 1:4 dilution in MenACWY group)] x 100. The combined VE across all strains was computed by mean of a generalized linear model; Test type: Other — Pre-specified; p = 0.0001, Generalized Linear Model; [statistical method as in outcome 1, analysis 1]; Vaccine Effectiveness = 51, 95% CI 2-sided [48 to 55]

3. Secondary Outcome: Percentages of Subjects Without Bactericidal Activity at 1:8 Dilution Against Each US N. Meningitidis Serogroup B Strain at 1 and 4 Months After the 3-dose Vaccination Series.
Description: The effectiveness of three doses of MenABCWY vaccine when compared to one dose of MenACWY vaccine against a panel of US N. meningitidis serogroup B invasive disease strains at 1 and 4 months after the 3-dose vaccination series were evaluated in terms of: the combined percentage of subjects without bactericidal activity at 1:8 dilution using the hSBA against each strain in MenABCWY Group and MenACWY Group. The data provided is an average of the percentage of subjects without bactericidal activity at 1:8 dilution across all 110 strains.
Time Frame: At Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Effectiveness (Months 7 & 10)- included all screened subjects who provided consent & demographic &/or baseline screening assessments, received subject ID & vaccination, & provided evaluable serum sample with the enc-hSBA result for at least 1 endemic N. meningitidis serogroup B invasive disease strain at Months 7 & 10.
Measure: Number; unit: Percentages of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 93 | 93
Percentages of subjects
  Combined Serogroup B Strains (Month 7) | 36.9 | 75.8
  Combined Serogroup B Strains (Month 10): number analyzed (Participants) | 90 | 90
  Combined Serogroup B Strains (Month 10) | 60.3 | 79.6
Statistical Analysis 1: Comparison: MenABCWY Group vs MenACWY Group; The Vaccine Effectiveness (VE) at 1 month after the 3-dose vaccination series for each strain is defined as [1 - (percentage of subjects without bactericidal activity at 1:8 dilution in MenABCWY group/percentage of subjects without bactericidal activity at 1:8 dilution in MenACWY group)] x 100. The combined VE across all strains was computed by mean of a generalized linear model; Test type: Other — Pre-specified; p = 0.0001, Generalized Linear Model; [statistical method as in outcome 1, analysis 1]; Vaccine Effectiveness = 51, 95% CI 2-sided [48 to 54]
Statistical Analysis 2: Comparison: MenABCWY Group vs MenACWY Group; The Vaccine Effectiveness (VE) at 4 months after the 3-dose vaccination series for each strain is defined as [1 - (percentage of subjects without bactericidal activity at 1:8 dilution in MenABCWY group/percentage of subjects without bactericidal activity at 1:8 dilution in MenACWY group)] x 100. The combined VE across all strains was computed by mean of a generalized linear model; Test type: Other — Pre-specified; p = 0.0001, Generalized Linear Model; [statistical method as in outcome 1, analysis 1]; Vaccine Effectiveness = 24, 95% CI [20 to 28]

4. Secondary Outcome: Percentages of US N. Meningitidis Serogroup B Strains Killed at 1:4 and 1:8 Dilutions at 1 and 4 Months After the 3-dose Vaccination Series
Description: The mean percentage of US N. meningitidis serogroup B strains killed by each subject, at 1:4 and 1:8 dilutions before the 3-dose vaccination series, at Month 6 (PRE) and at 1 and 4 months after the 3-dose vaccination series (Month 7 and Month 10).
Time Frame: At Month 6 (before the 3-dose vaccination series) and at Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Effectiveness (Months 6, 7 & 10)- included all screened subjects who provided consent & demographic &/or baseline screening assessments, got subject ID & vaccination, & provided serum sample with enc-hSBA result for at least 1 endemic N. meningitidis serogroup B invasive disease strain before Month 6 & at Months 7 & 10
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 93 | 93
Percentage
  1:4, PRE | 56.97 (18.134) | 22.94 (17.764)
  1:4, Month 7 | 77.78 (10.041) | 21.91 (16.885)
  1:4, Month 10: number analyzed (Participants) | 90 | 90
  1:4, Month 10 | 62.37 (15.976) | 22.49 (17.094)
  1:8, PRE | 28.81 (17.086) | 11.53 (11.705)
  1:8, Month 7 | 56.95 (14.389) | 11.4 (11.266)
  1:8, Month 10: number analyzed (Participants) | 90 | 90
  1:8, Month 10 | 31.46 (19.434) | 11.15 (10.774)

5. Secondary Outcome: Percentages of Subjects With Enc-hSBA ≥ 1:4 and Enc-hSBA ≥1:8 at 1 and 4 Months After the 3-dose Vaccination Series
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY vaccine, in terms of percentages of subjects with enc-hSBA ≥ 1:4 and enc-hSBA ≥ 1:8 against four N. meningitidis serogroup B test strains (M14459, M07-0241084, 96217 and NZ98/254) at 1 and 4 months after the 3-dose vaccination series (Month 7 and Month 10).
Time Frame: At Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Immunogenicity (Months 7 &10)- included all screened subjects who provided consent & demographic &/or baseline screening assessments, received a subject ID & vaccination, & provided evaluable serum samples at Months 7 & 10 & whose immunogenicity assay result was available for at least one serogroup B test strain.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 92 | 91
Percentages of subjects
  M14459 (≥ 1:4, Month 7): number analyzed (Participants) | 91 | 90
  M14459 (≥ 1:4, Month 7) | 98 [92.3 to 99.73] | 12 [6.3 to 20.8]
  M14459 (≥ 1:4, Month 10): number analyzed (Participants) | 87 | 90
  M14459 (≥ 1:4, Month 10) | 72 [61.8 to 81.5] | 12 [6.3 to 20.8]
  M14459 (≥ 1:8, Month 7): number analyzed (Participants) | 91 | 90
  M14459 (≥ 1:8, Month 7) | 67 [56.4 to 76.5] | 2 [0.27 to 7.8]
  M14459 (≥ 1:8, Month 10): number analyzed (Participants) | 87 | 90
  M14459 (≥ 1:8, Month 10) | 21 [12.7 to 30.7] | 1 [0.03 to 6]
  M07-0241084 (≥ 1:4, Month 7): number analyzed (Participants) | 90 | 85
  M07-0241084 (≥ 1:4, Month 7) | 81 [71.5 to 88.6] | 21 [13.1 to 31.4]
  M07-0241084 (≥ 1:4, Month 10): number analyzed (Participants) | 79 | 78
  M07-0241084 (≥ 1:4, Month 10) | 46 [34.3 to 57.2] | 22 [13.2 to 32.6]
  M07-0241084 (≥ 1:8, Month 7): number analyzed (Participants) | 90 | 85
  M07-0241084 (≥ 1:8, Month 7) | 38 [27.8 to 48.6] | 5 [1.3 to 11.6]
  M07-0241084 (≥ 1:8, Month 10): number analyzed (Participants) | 79 | 78
  M07-0241084 (≥ 1:8, Month 10) | 11 [5.3 to 20.5] | 6 [2.1 to 14.3]
  96217 (≥ 1:4, Month 7): number analyzed (Participants) | 89 | 88
  96217 (≥ 1:4, Month 7) | 99 [93.9 to 99.97] | 48 [37 to 58.6]
  96217 (≥ 1:4, Month 10): number analyzed (Participants) | 87 | 88
  96217 (≥ 1:4, Month 10) | 100 [95.8 to 100] | 41 [30.5 to 51.9]
  96217 (≥ 1:8, Month 7): number analyzed (Participants) | 89 | 88
  96217 (≥ 1:8, Month 7) | 99 [93.9 to 99.97] | 17 [9.9 to 26.6]
  96217 (≥ 1:8, Month 10): number analyzed (Participants) | 87 | 88
  96217 (≥ 1:8, Month 10) | 99 [93.8 to 99.97] | 16 [9 to 25.2]
  NZ98/254 (≥ 1:4, Month 7): number analyzed (Participants) | 84 | 87
  NZ98/254 (≥ 1:4, Month 7) | 76 [65.7 to 84.8] | 1 [0.03 to 6.2]
  NZ98/254 (≥ 1:4, Month 10): number analyzed (Participants) | 80 | 83
  NZ98/254 (≥ 1:4, Month 10) | 34 [23.6 to 45.2] | 1 [0.03 to 6.5]
  NZ98/254 (≥ 1:8, Month 7): number analyzed (Participants) | 84 | 87
  NZ98/254 (≥ 1:8, Month 7) | 39 [28.8 to 50.5] | 1 [0.03 to 6.2]
  NZ98/254 (≥ 1:8, Month 10): number analyzed (Participants) | 80 | 83
  NZ98/254 (≥ 1:8, Month 10) | 4 [0.8 to 10.6] | 0 [0 to 4.3]

6. Secondary Outcome: HT-hSBA Geometric Mean Titers (GMTs) Against the N. Meningitidis Serogroup B Test Strains
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY vaccine, in terms of HT-hSBA GMTs against four N. meningitidis serogroup B test strains (M14459, M07-0241084, 96217 and NZ98/254) after the 3-dose vaccination series.
Time Frame: At Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 91 | 91
Titers
  M14459, Month 7: number analyzed (Participants) | 91 | 88
  M14459, Month 7 | 23.12 [20 to 27] | 1.1 [0.94 to 1.29]
  M14459, Month 10: number analyzed (Participants) | 88 | 91
  M14459, Month 10 | 3.93 [3.14 to 4.91] | 1.18 [0.95 to 1.46]
  M07-0241084, Month 7: number analyzed (Participants) | 89 | 90
  M07-0241084, Month 7 | 12.26 [9.59 to 16] | 1.74 [1.37 to 2.2]
  M07-0241084, Month 10: number analyzed (Participants) | 86 | 90
  M07-0241084, Month 10 | 3.04 [2.36 to 3.92] | 1.68 [1.31 to 2.14]
  96217, Month 7: number analyzed (Participants) | 90 | 87
  96217, Month 7 | 367.29 [277 to 486] | 4.02 [3.03 to 5.32]
  96217, Month 10: number analyzed (Participants) | 87 | 85
  96217, Month 10 | 142.06 [105 to 191] | 3.32 [2.46 to 4.48]
  NZ98/254, Month 7: number analyzed (Participants) | 89 | 89
  NZ98/254, Month 7 | 19.69 [16 to 24] | 1.02 [0.85 to 1.23]
  NZ98/254, Month 10: number analyzed (Participants) | 87 | 90
  NZ98/254, Month 10 | 3.75 [3.01 to 4.68] | 1.04 [0.84 to 1.29]

7. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against N. Meningitidis Serogroup B Test Strains ≥ Lower Limit of Quantitation (LLQ) at 1 Month After the 3-dose Vaccination Series.
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of percentages of subjects with HT-hSBA titers ≥ LLQ against serogroup N. meningitidis B test strains (M14459, M07-0241084, 96217 and NZ98/254), at 1 month after the 3-dose vaccination series.The LLQ cut off values for strains 96217, M07-0241084,M14459 and NZ98/254 were 8.6, 8.9, 8 and 8.2 respectively.
Time Frame: At Month 7 (1 month after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Immunogenicity (Month 7)- included all screened subjects who provided consent & demographic &/or baseline screening assessments, received a subject ID & vaccination, & provided evaluable serum samples at Month 7 & whose immunogenicity assay result was available for at least one serogroup B test strain.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 91 | 90
Percentages of subjects
  M07-0241084, Month 7: number analyzed (Participants) | 89 | 90
  M07-0241084, Month 7 | 63 [52.0 to 72.9] | 12 [6.3 to 20.8]
  M14459, Month 7: number analyzed (Participants) | 91 | 88
  M14459, Month 7 | 90 [82.1 to 95.4] | 1 [0.03 to 6.2]
  NZ98/254, Month 7: number analyzed (Participants) | 89 | 89
  NZ98/254, Month 7 | 79 [68.7 to 86.6] | 1 [0.03 to 6.1]
  96217, Month 7: number analyzed (Participants) | 90 | 87
  96217, Month 7 | 100 [96.0 to 100.0] | 37 [26.7 to 47.8]

8. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against N. Meningitidis Serogroup B Test Strains ≥ LLQ at 4 Months After the 3-dose Vaccination Series
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of percentages of subjects with HT-hSBA titers ≥ LLQ against serogroup N. meningitidis B test strains (M14459, M07-0241084, 96217 and NZ98/254), at 4 months after the 3-dose vaccination series.
  The LLQ cut off values for the strains 96217, M07-0241084,M14459 and NZ98/254 were 8.6,8.9, 8 and 8.2 respectively.
Time Frame: At Month 10 (4 months after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Immunogenicity (Month 10)- included all screened subjects who provided informed consent & demographic &/or baseline screening assessments, received a subject ID & vaccination, & provided evaluable serum samples at Month 10 and whose immunogenicity assay result was available for at least one serogroup strain.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 88 | 91
Percentages of subjects
  96217: number analyzed (Participants) | 87 | 85
  96217 | 99 [93.8 to 99.97] | 32 [22.1 to 42.8]
  M07-0241084: number analyzed (Participants) | 86 | 90
  M07-0241084 | 23 [14.8 to 33.6] | 12 [6.3 to 20.8]
  M14459 | 36 [26.4 to 47.3] | 3 [0.7 to 9.3]
  NZ98/254: number analyzed (Participants) | 87 | 90
  NZ98/254 | 33 [23.6 to 44.3] | 1 [0.03 to 6.0]

9. Secondary Outcome: Percentages of Subjects With a Two-fold Rise in HT-hSBA Titers Against the N. Meningitidis Serogroup B Test Strains at 1 and 4 Months After the 3-dose Vaccination Series.
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a two-fold rise in HT-hSBA titers against the N. meningitidis serogroup B test strains, at 1 and 4 months after the 3-dose vaccination series. The two-fold titers rise is defined as: a) for subjects with pre-vaccination (month 6 from the parent study) HT-hSBA titers < LLQ, postvaccination HT-hSBA titers ≥ 2 LLQ; b) for subjects with pre-vaccination (month 6 from the parent study) HT-hSBA titers ≥ LLQ, an increase of at least two times the pre-vaccination HT-hSBA titers.
Time Frame: At Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: Analysis was performed on the FAS-Immunogenicity (months 7 and 10)- included all screened subjects who provided consent & demographic &/baseline screening assessments, received a subjects D & vaccination, & provided evaluable serum samples at months 7 & 10 & whose immunogenicity assay result was available for at least one serogroup B strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 90 | 90
Percentage of subjects
  96217 (Month 7): number analyzed (Participants) | 87 | 86
  96217 (Month 7) | 87 [78.5 to 93.5] | 12 [5.7 to 20.4]
  M07-0241084 (Month 7): number analyzed (Participants) | 84 | 85
  M07-0241084 (Month 7) | 38 [27.7 to 49.3] | 1 [0.03 to 6.4]
  M14459 (Month 7): number analyzed (Participants) | 90 | 87
  M14459 (Month 7) | 67 [56.0 to 76.3] | 0 [0 to 4.1]
  NZ98/254 (Month 7): number analyzed (Participants) | 88 | 88
  NZ98/254 (Month 7) | 56 [44.7 to 66.3] | 0 [0 to 4.1]
  96217 (Month 10): number analyzed (Participants) | 84 | 84
  96217 (Month 10) | 54 [42.4 to 64.5] | 7 [2.7 to 14.9]
  M07-0241084 (Month 10): number analyzed (Participants) | 81 | 85
  M07-0241084 (Month 10) | 0 [0 to 4.4] | 4 [0.7 to 10.0]
  M14459 (Month 10): number analyzed (Participants) | 87 | 90
  M14459 (Month 10) | 7 [2.6 to 14.4] | 0 [0 to 4]
  NZ98/254 (Month 10): number analyzed (Participants) | 86 | 89
  NZ98/254 (Month 10) | 13 [6.6 to 21.7] | 0 [0 to 4.1]

10. Secondary Outcome: Percentages of Subjects With a Three-fold Rise in HT-hSBA Titers Against the N. Meningitidis Serogroup B Test Strains at 1 and 4 Months After the 3-dose Vaccination Series.
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a three-fold rise in HT-hSBA titers against the N. meningitidis serogroup B test strains, at 1 and 4 months after the 3-dose vaccination series. The three-fold titers rise is defined as: a) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers < LLQ, postvaccination HT-hSBA titers ≥ 3 LLQ; b) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers ≥ LLQ, an increase of at least three times the pre-vaccination HT-hSBA titers.
Time Frame: At months 7 and 10 (1 and 4 months after 3-dose vaccination series)
Population: Analysis was performed on the FAS-Immunogenicity (months 7 and 10)- included all screened subjects who provided consent & demographic &/baseline screening assessments, received a subject ID & vaccination, & provided evaluable serum samples at months 7 & 10 & whose immunogenicity assay result was available for at least one serogroup B strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 90 | 90
Percentage of subjects
  96217 (Month 7): number analyzed (Participants) | 87 | 86
  96217 (Month 7) | 79 [69.3 to 87.3] | 5 [1.3 to 11.5]
  M07-0241084 (Month 7): number analyzed (Participants) | 84 | 85
  M07-0241084 (Month 7) | 23 [14.2 to 33.1] | 1 [0.03 to 6.4]
  M14459 (Month 7): number analyzed (Participants) | 90 | 87
  M14459 (Month 7) | 41 [30.8 to 52.0] | 0 [0 to 4.1]
  NZ98/254 (Month 7): number analyzed (Participants) | 88 | 88
  NZ98/254 (Month 7) | 41 [30.5 to 51.9] | 0 [0 to 4.1]
  96217 (Month 10): number analyzed (Participants) | 84 | 84
  96217 (Month 10) | 27 [18.2 to 38.2] | 5 [1.3 to 11.8]
  M07-0241084 (Month 10): number analyzed (Participants) | 81 | 85
  M07-0241084 (Month 10) | 0 [0 to 4.4] | 2 [0.29 to 8.2]
  M14459 (Month 10): number analyzed (Participants) | 87 | 90
  M14459 (Month 10) | 3 [0.7 to 9.8] | 0 [0 to 4]
  NZ98/254 (Month 10): number analyzed (Participants) | 86 | 89
  NZ98/254 (Month 10) | 5 [1.3 to 11.5] | 0 [0 to 4.1]

11. Secondary Outcome: Percentages of Subjects With a Four-fold Rise in HT-hSBA Titers Against the N. Meningitidis Serogroup B Test Strains at 1 and 4 Months After the 3-dose Vaccination Series.
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a four-fold rise in HT-hSBA titers against the N. meningitidis serogroup B test strains, at 1 and 4 months after the 3-dose vaccination series. The four-fold titers rise is defined as: a) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers < LLQ, postvaccination HT-hSBA titers ≥ 4 LLQ; b) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers ≥ LLQ, an increase of at least four times the pre-vaccination HT-hSBA titers.
Time Frame: At Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 90 | 90
Percentages of subjects
  96217 (Month 7): number analyzed (Participants) | 87 | 86
  96217 (Month 7) | 63 [52.2 to 73.3] | 3 [0.7 to 9.9]
  M07-0241084 (Month 7): number analyzed (Participants) | 84 | 85
  M07-0241084 (Month 7) | 12 [5.9 to 20.8] | 0 [0 to 4.2]
  M14459 (Month 7): number analyzed (Participants) | 90 | 87
  M14459 (Month 7) | 23 [15.1 to 33.4] | 0 [0.0 to 4.1]
  NZ98/254 (Month 7): number analyzed (Participants) | 88 | 88
  NZ98/254 (Month 7) | 33 [23.3 to 43.8] | 0 [0.0 to 4.1]
  96217 (Month 10): number analyzed (Participants) | 84 | 84
  96217 (Month 10) | 15 [8.5 to 25.0] | 5 [1.3 to 11.8]
  M07-0241084 (Month 10): number analyzed (Participants) | 81 | 85
  M07-0241084 (Month 10) | 0 [0 to 4.4] | 1 [0.03 to 6.4]
  M14459 (Month 10): number analyzed (Participants) | 87 | 90
  M14459 (Month 10) | 3 [0.7 to 9.8] | 0 [0 to 4]
  NZ98/254 (Month 10): number analyzed (Participants) | 86 | 89
  NZ98/254 (Month 10) | 2 [0.28 to 8.2] | 0 [0 to 4.1]

12. Secondary Outcome: HT-hSBA GMTs Against N. Meningitidis Serogroups A, C, W and Y.
Description: The immunogenicity of three doses of MenABCWY compared to a single dose of MenACWY vaccine, in terms of HT-hSBA GMTs to serogroups A, C, W, and Y, at 1 and 4 months after the 3-dose vaccination series.
Time Frame: At Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 91 | 91
Titers
  Men A, Month 7: number analyzed (Participants) | 91 | 87
  Men A, Month 7 | 127.92 [91 to 179] | 3.37 [2.41 to 4.73]
  Men A, Month 10: number analyzed (Participants) | 85 | 88
  Men A, Month 10 | 36.5 [25 to 53] | 2.73 [1.89 to 3.94]
  Men C, Month 7: number analyzed (Participants) | 85 | 86
  Men C, Month 7 | 521.64 [365 to 745] | 18.34 [13 to 26]
  Men C, Month 10: number analyzed (Participants) | 86 | 89
  Men C, Month 10 | 291.19 [201 to 421] | 15.4 [11 to 22]
  Men W, Month 7: number analyzed (Participants) | 83 | 88
  Men W, Month 7 | 424.8 [310 to 581] | 40.22 [30 to 54]
  Men W, Month 10: number analyzed (Participants) | 85 | 83
  Men W, Month 10 | 147.4 [104 to 209] | 23.01 [16 to 33]
  Men Y, Month 7: number analyzed (Participants) | 91 | 88
  Men Y, Month 7 | 204.84 [142 to 296] | 13.27 [9.21 to 19]
  Men Y, Month 10: number analyzed (Participants) | 86 | 91
  Men Y, Month 10 | 83.42 [55 to 126] | 11.85 [7.93 to 18]

13. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against the N. Meningitidis Serogroup A, C, W and Y ≥ LLQ at 1 Month After the 3- Dose Vaccination Series
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers ≥ LLQ against serogroups A, C, W, Y, at 1 month after the 3-dose vaccination series.The LLQ cut off values for serogroups A,C,W and Y were 22.7,5.2, 39.6 and 14.7 respectively.
Time Frame: At Month 7 (1 month after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Immunogenicity (Month 7)- included all screened subjects who provided consent & demographic &/or baseline screening assessments, received a subject ID & vaccination, & provided evaluable serum samples at Month 7 & whose immunogenicity assay result was available for at least one serogroup A, C, W and Y test strain.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 91 | 88
Percentages of subjects
  Men A: number analyzed (Participants) | 91 | 87
  Men A | 98 [92.3 to 99.73] | 24 [15.6 to 34.5]
  Men C: number analyzed (Participants) | 85 | 86
  Men C | 100 [95.8 to 100.0] | 73 [62.6 to 82.2]
  Men W: number analyzed (Participants) | 83 | 88
  Men W | 99 [93.5 to 99.97] | 60 [49.2 to 70.5]
  Men Y | 100 [96.0 to 100] | 57 [45.8 to 67.3]

14. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against the N. Meningitidis Serogroup A, C, W and Y ≥ LLQ at 4 Months After the 3-dose Vaccination Series
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers ≥ LLQ against serogroups A, C, W, Y, at 4 months after the 3-dose vaccination series. The LLQ cut off values for serogroups A, C, W and Y were 22.7,5.2,39.6 and 14.7 respectively.
Time Frame: At Month 10 (4 months after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Immunogenicity (Month 10)- included all screened subjects who provided informed consent & demographic &/or baseline screening assessments, received a subject ID & vaccination, & provided evaluable serum samples at Month 10 and whose immunogenicity assay result was available for at least one serogroup B strain
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 86 | 91
Percentages of subjects
  Men A: number analyzed (Participants) | 85 | 88
  Men A | 81 [71.2 to 88.8] | 18 [10.8 to 27.8]
  Men C: number analyzed (Participants) | 86 | 89
  Men C | 100 [95.8 to 100.0] | 69 [57.8 to 78.0]
  Men W: number analyzed (Participants) | 85 | 83
  Men W | 89 [80.9 to 95.0] | 51 [39.4 to 61.8]
  Men Y | 86 [76.9 to 92.6] | 53 [42.0 to 63.3]

15. Secondary Outcome: Percentage of Subjects With Two-fold Rise in HT-hSBA Titers Against the N. Meningitidis Serogroups A, C,W and Y at 1 and 4 Months After the 3-dose Vaccination Series.
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a two-fold rise in HT-hSBA titers against the N. meningitidis serogroups A, C, W and Y at 1 and 4 months after the 3-dose vaccination series. The two-fold titers rise is defined as: a) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers < LLQ, postvaccination HT-hSBA titers ≥ 2 LLQ; b) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers ≥ LLQ, an increase of at least two times the pre-vaccination HT-hSBA titers.
Time Frame: At Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 89 | 88
Percentage of subjects
  Men A, Month 7: number analyzed (Participants) | 83 | 85
  Men A, Month 7 | 88 [79.0 to 94.1] | 2 [0.29 to 8.2]
  Men C, Month 7: number analyzed (Participants) | 84 | 84
  Men C, Month 7 | 87 [77.8 to 93.3] | 2 [0.29 to 8.3]
  Men W, Month 7: number analyzed (Participants) | 81 | 84
  Men W, Month 7 | 83 [72.7 to 90.2] | 5 [1.3 to 11.8]
  Men Y, Month 7: number analyzed (Participants) | 89 | 85
  Men Y, Month 7 | 57 [46.4 to 67.7] | 2 [0.29 to 8.2]
  Men A, Month 10: number analyzed (Participants) | 77 | 86
  Men A, Month 10 | 32 [22.2 to 44.1] | 1 [0.03 to 6.3]
  Men C, Month 10: number analyzed (Participants) | 85 | 87
  Men C, Month 10 | 56 [45.3 to 67.2] | 8 [3.3 to 15.9]
  Men W, Month 10: number analyzed (Participants) | 83 | 79
  Men W, Month 10 | 24 [15.4 to 34.7] | 1 [0.03 to 6.9]
  Men Y, Month 10: number analyzed (Participants) | 84 | 88
  Men Y, Month 10 | 26 [17.2 to 36.9] | 3 [0.7 to 9.6]

16. Secondary Outcome: Percentage of Subjects With Three-fold Rise in HT-hSBA Titers Against the N. Meningitidis Serogroups A, C, W and Y at 1 and 4 Months After the 3-dose Vaccination Series.
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a three-fold rise in HT-hSBA titers against the N. meningitidis serogroups A, C, W and Y, at 1 and 4 months after the 3-dose vaccination series. The three-fold titers rise is defined as: a) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers < LLQ, postvaccination HT-hSBA titers ≥ 3 LLQ; b) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers ≥ LLQ, an increase of at least three times the pre-vaccination HT-hSBA titers.
Time Frame: At Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 89 | 88
Percentage of subjects
  Men A, Month 7: number analyzed (Participants) | 83 | 85
  Men A, Month 7 | 69 [57.6 to 78.4] | 0 [0 to 4.2]
  Men C, Month 7: number analyzed (Participants) | 84 | 84
  Men C, Month 7 | 60 [48.3 to 70.1] | 1 [0.03 to 6.5]
  Men W, Month 7: number analyzed (Participants) | 81 | 84
  Men W, Month 7 | 67 [55.3 to 76.8] | 0 [0 to 4.3]
  Men Y, Month 7: number analyzed (Participants) | 89 | 85
  Men Y, Month 7 | 39 [29.1 to 50.3] | 0 [0 to 4.2]
  Men A, Month 10: number analyzed (Participants) | 77 | 86
  Men A, Month 10 | 16 [8.3 to 25.6] | 1 [0.03 to 6.3]
  Men C, Month 10: number analyzed (Participants) | 85 | 87
  Men C, Month 10 | 29 [20.0 to 40.3] | 5 [1.3 to 11.4]
  Men W, Month 10: number analyzed (Participants) | 83 | 79
  Men W, Month 10 | 13 [6.8 to 22.5] | 0 [0 to 4.6]
  Men Y, Month 10: number analyzed (Participants) | 84 | 88
  Men Y, Month 10 | 15 [8.5 to 25.0] | 2 [0.28 to 8.0]

17. Secondary Outcome: Percentage of Subjects With Four-fold Rise in HT-hSBA Titers Against the N. Meningitidis Serogroups A, C, W and Y at 1 and 4 Months After the 3-dose Vaccination Series.
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a four-fold rise in HT-hSBA titers against the N. meningitidis serogroups A, C, W and Y, at 1 and 4 months after the 3-dose vaccination series. The four-fold titers rise is defined as: a) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers < LLQ, postvaccination HT-hSBA titers ≥ 4 LLQ; b) for subjects with pre-vaccination (Month 6 from the parent study) HT-hSBA titers ≥ LLQ, an increase of at least four times the pre-vaccination HT-hSBA titers.
Time Frame: At Months 7 and 10 (1 and 4 months after the 3-dose vaccination series)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 89 | 88
Percentage of subjects
  Men A, Month 7: number analyzed (Participants) | 83 | 85
  Men A, Month 7 | 53 [41.7 to 64.1] | 0 [0 to 4.2]
  Men C, Month 7: number analyzed (Participants) | 84 | 84
  Men C, Month 7 | 49 [37.7 to 60.0] | 1 [0.03 to 6.5]
  Men W, Month 7: number analyzed (Participants) | 81 | 84
  Men W, Month 7 | 49 [38.1 to 60.7] | 0 [0 to 4.3]
  Men Y, Month 7: number analyzed (Participants) | 89 | 85
  Men Y, Month 7 | 28 [19.1 to 38.6] | 0 [0 to 4.2]
  Men A, Month 10: number analyzed (Participants) | 77 | 86
  Men A, Month 10 | 6 [2.1 to 14.5] | 1 [0.03 to 6.3]
  Men C, Month 10: number analyzed (Participants) | 85 | 87
  Men C, Month 10 | 21 [13.1 to 31.4] | 2 [0.28 to 8.1]
  Men W, Month 10: number analyzed (Participants) | 83 | 79
  Men W, Month 10 | 8 [3.5 to 16.6] | 0 [0 to 4.6]
  Men Y, Month 10: number analyzed (Participants) | 84 | 88
  Men Y, Month 10 | 6 [2.0 to 13.4] | 1 [0.03 to 6.2]

18. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against N. Meningitidis Serogroup B Test Strains≥ 5, ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 at 1 Month After the 3-dose Vaccination Series
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of percentages of subjects with HT-hSBA titers ≥ 5, ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 against serogroup N. meningitidis B test strains (M14459, M07-0241084, 96217 and NZ98/254), at 1 month after the 3-dose vaccination series.
Time Frame: At Month 7 (1 month after the 3-dose vaccination series)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 91 | 90
Percentage of subjects
  96217, ≥ 5: number analyzed (Participants) | 90 | 87
  96217, ≥ 5 | 100 [96 to 100] | 38 [27.7 to 49]
  96217, ≥ 8: number analyzed (Participants) | 90 | 87
  96217, ≥ 8 | 100 [96 to 100] | 37 [26.7 to 47.8]
  96217, ≥ 16: number analyzed (Participants) | 90 | 87
  96217, ≥ 16 | 100 [96 to 100] | 25 [16.6 to 35.7]
  96217, ≥ 32: number analyzed (Participants) | 90 | 87
  96217, ≥ 32 | 100 [96 to 100] | 15 [8.2 to 24.2]
  96217, ≥ 64: number analyzed (Participants) | 90 | 87
  96217, ≥ 64 | 99 [94 to 99.97] | 8 [3.3 to 15.9]
  96217, ≥ 128: number analyzed (Participants) | 90 | 87
  96217, ≥ 128 | 93 [86.1 to 97.5] | 3 [0.7 to 9.7]
  M07-0241084, ≥ 5: number analyzed (Participants) | 89 | 90
  M07-0241084, ≥ 5 | 82 [72.5 to 89.4] | 16 [8.8 to 24.7]
  M07-0241084, ≥ 8: number analyzed (Participants) | 89 | 90
  M07-0241084, ≥ 8 | 67 [56.7 to 77] | 12 [6.3 to 20.8]
  M07-0241084, ≥ 16: number analyzed (Participants) | 89 | 90
  M07-0241084, ≥ 16 | 46 [35.4 to 57] | 8 [3.2 to 15.4]
  M07-0241084, ≥ 32: number analyzed (Participants) | 89 | 90
  M07-0241084, ≥ 32 | 20 [12.4 to 30.1] | 3 [0.7 to 9.4]
  M07-0241084, ≥ 64: number analyzed (Participants) | 89 | 90
  M07-0241084, ≥ 64 | 6 [1.8 to 12.6] | 2 [0.27 to 7.8]
  M07-0241084, ≥ 128: number analyzed (Participants) | 89 | 90
  M07-0241084, ≥ 128 | 0 [0 to 4.1] | 0 [0 to 4]
  M14459, ≥ 5: number analyzed (Participants) | 91 | 88
  M14459, ≥ 5 | 95 [87.6 to 98.2] | 1 [0.03 to 6.2]
  M14459, ≥ 8: number analyzed (Participants) | 91 | 88
  M14459, ≥ 8 | 90 [82.1 to 95.4] | 1 [0.03 to 6.2]
  M14459, ≥ 16: number analyzed (Participants) | 91 | 88
  M14459, ≥ 16 | 71 [61 to 80.4] | 1 [0.03 to 6.2]
  M14459, ≥ 32: number analyzed (Participants) | 91 | 88
  M14459, ≥ 32 | 34 [24.5 to 44.7] | 1 [0.03 to 6.2]
  M14459, ≥ 64: number analyzed (Participants) | 91 | 88
  M14459, ≥ 64 | 11 [5.4 to 19.3] | 0 [0 to 4.1]
  M14459, ≥ 128: number analyzed (Participants) | 91 | 88
  M14459, ≥ 128 | 3 [0.7 to 9.3] | 0 [0 to 4.1]
  NZ98/254, ≥ 5: number analyzed (Participants) | 89 | 89
  NZ98/254, ≥ 5 | 89 [80.3 to 94.5] | 1 [0.03 to 6.1]
  NZ98/254, ≥ 8: number analyzed (Participants) | 89 | 89
  NZ98/254, ≥ 8 | 79 [68.7 to 86.6] | 1 [0.03 to 6.1]
  NZ98/254, ≥ 16: number analyzed (Participants) | 89 | 89
  NZ98/254, ≥ 16 | 61 [49.7 to 70.9] | 0 [0 to 4.1]
  NZ98/254, ≥ 32: number analyzed (Participants) | 89 | 89
  NZ98/254, ≥ 32 | 37 [27.1 to 48] | 0 [0 to 4.1]
  NZ98/254, ≥ 64: number analyzed (Participants) | 89 | 89
  NZ98/254, ≥ 64 | 10 [4.7 to 18.3] | 0 [0 to 4.1]
  NZ98/254, ≥ 128: number analyzed (Participants) | 89 | 89
  NZ98/254, ≥ 128 | 4 [1.2 to 11.1] | 0 [0 to 4.1]

19. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against N. Meningitidis Serogroup B Test Strains ≥ 5, ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 at 4 Months After the 3-dose Vaccination Series
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of percentages of subjects with HT-hSBA titers ≥ 5, ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 against serogroup N. meningitidis B test strains (M14459, M07-0241084, 96217 and NZ98/254), at 4 months after the 3-dose vaccination series.
Time Frame: At Month 10 (4 months after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Immunogenicity (Month 10)- included all screened subjects who provided consent & demographic &/or baseline screening assessments, received a subject ID & vaccination, & provided evaluable serum samples at Month 10 & whose immunogenicity assay result was available for at least one serogroup B test strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 88 | 91
Percentage of subjects
  96217, ≥ 5: number analyzed (Participants) | 87 | 85
  96217, ≥ 5 | 99 [93.8 to 99.97] | 35 [25.2 to 46.4]
  96217, ≥ 8: number analyzed (Participants) | 87 | 85
  96217, ≥ 8 | 99 [93.8 to 99.97] | 33 [23.1 to 44]
  96217, ≥ 16: number analyzed (Participants) | 87 | 85
  96217, ≥ 16 | 98 [91.9 to 99.72] | 21 [13.1 to 31.4]
  96217, ≥ 32: number analyzed (Participants) | 87 | 85
  96217, ≥ 32 | 94 [87.1 to 98.1] | 16 [9.3 to 26.1]
  96217, ≥ 64: number analyzed (Participants) | 87 | 85
  96217, ≥ 64 | 85 [75.8 to 91.8] | 6 [1.9 to 13.2]
  96217, ≥ 128: number analyzed (Participants) | 87 | 85
  96217, ≥ 128 | 56 [45.3 to 66.9] | 2 [0.29 to 8.2]
  M07-0241084, ≥ 5: number analyzed (Participants) | 86 | 90
  M07-0241084, ≥ 5 | 38 [28.1 to 49.5] | 17 [9.6 to 26]
  M07-0241084, ≥ 8: number analyzed (Participants) | 86 | 90
  M07-0241084, ≥ 8 | 24 [15.8 to 34.9] | 12 [6.3 to 20.8]
  M07-0241084, ≥ 16: number analyzed (Participants) | 86 | 90
  M07-0241084, ≥ 16 | 9 [4.1 to 17.5] | 9 [3.9 to 16.8]
  M07-0241084, ≥ 32: number analyzed (Participants) | 86 | 90
  M07-0241084, ≥ 32 | 1 [0.03 to 6.3] | 3 [0.7 to 9.4]
  M07-0241084, ≥ 64: number analyzed (Participants) | 86 | 90
  M07-0241084, ≥ 64 | 1 [0.03 to 6.3] | 2 [0.27 to 7.8]
  M07-0241084, ≥ 128: number analyzed (Participants) | 86 | 90
  M07-0241084, ≥ 128 | 0 [0 to 4.2] | 1 [0.03 to 6]
  M14459, ≥ 5 | 49 [38.1 to 59.8] | 4 [1.2 to 10.9]
  M14459, ≥ 8 | 36 [26.4 to 47.3] | 3 [0.7 to 9.3]
  M14459, ≥ 16 | 17 [9.9 to 26.6] | 1 [0.03 to 6]
  M14459, ≥ 32 | 6 [1.9 to 12.8] | 0 [0 to 4]
  M14459, ≥ 64 | 1 [0.03 to 6.2] | 0 [0 to 4]
  M14459, ≥ 128 | 0 [0 to 4.1] | 0 [0 to 4]
  NZ98/254, ≥ 5: number analyzed (Participants) | 87 | 90
  NZ98/254, ≥ 5 | 44 [33.1 to 54.7] | 1 [0.03 to 6]
  NZ98/254, ≥ 8: number analyzed (Participants) | 87 | 90
  NZ98/254, ≥ 8 | 34 [24.6 to 45.4] | 1 [0.03 to 6]
  NZ98/254, ≥ 16: number analyzed (Participants) | 87 | 90
  NZ98/254, ≥ 16 | 16 [9.1 to 25.5] | 0 [0 to 4]
  NZ98/254, ≥ 32: number analyzed (Participants) | 87 | 90
  NZ98/254, ≥ 32 | 5 [1.3 to 11.4] | 0 [0 to 4]
  NZ98/254, ≥ 64: number analyzed (Participants) | 87 | 90
  NZ98/254, ≥ 64 | 2 [0.28 to 8.1] | 0 [0 to 4]
  NZ98/254, ≥ 128: number analyzed (Participants) | 87 | 90
  NZ98/254, ≥ 128 | 2 [0.28 to 8.1] | 0 [0 to 4]

20. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against the N. Meningitidis Serogroup A, C, W and Y ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥128 at 1 Month After the 3- Dose Vaccination Series
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥128 against serogroups A, C, W, Y, at 1 month after the 3-dose vaccination series.
Time Frame: At Month 7 (1 month after the 3-dose vaccination series)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 91 | 88
Percentage of subjects
  Men A, ≥ 8: number analyzed (Participants) | 91 | 87
  Men A, ≥ 8 | 98 [92.3 to 99.73] | 30 [20.5 to 40.6]
  Men A, ≥ 16: number analyzed (Participants) | 91 | 87
  Men A, ≥ 16 | 98 [92.3 to 99.73] | 26 [17.6 to 37]
  Men A, ≥ 32 | 98 [92.3 to 99.73] | 22 [13.7 to 32]
  Men A, ≥ 64: number analyzed (Participants) | 91 | 87
  Men A, ≥ 64 | 86 [76.8 to 92.2] | 13 [6.5 to 21.5]
  Men A, ≥ 128: number analyzed (Participants) | 91 | 87
  Men A, ≥ 128 | 56 [45.2 to 66.4] | 8 [3.3 to 15.9]
  Men C, ≥ 8: number analyzed (Participants) | 85 | 86
  Men C, ≥ 8 | 100 [95.8 to 100] | 71 [60.1 to 80.2]
  Men C, ≥ 16: number analyzed (Participants) | 85 | 86
  Men C, ≥ 16 | 99 [93.6 to 99.97] | 51 [40.1 to 62.1]
  Men C, ≥ 32: number analyzed (Participants) | 85 | 86
  Men C, ≥ 32 | 99 [93.6 to 99.97] | 33 [22.8 to 43.5]
  Men C, ≥ 64: number analyzed (Participants) | 85 | 86
  Men C, ≥ 64 | 99 [93.6 to 99.97] | 26 [16.8 to 36.1]
  Men C, ≥ 128: number analyzed (Participants) | 85 | 86
  Men C, ≥ 128 | 91 [82.3 to 95.8] | 19 [11 to 28.4]
  Men W, ≥ 8: number analyzed (Participants) | 83 | 88
  Men W, ≥ 8 | 100 [95.7 to 100] | 86 [77.4 to 92.8]
  Men W, ≥ 16: number analyzed (Participants) | 83 | 88
  Men W, ≥ 16 | 100 [95.7 to 100] | 77 [67.1 to 85.5]
  Men W, ≥ 32: number analyzed (Participants) | 83 | 88
  Men W, ≥ 32 | 99 [93.5 to 99.97] | 61 [50.4 to 71.6]
  Men W, ≥ 64: number analyzed (Participants) | 83 | 88
  Men W, ≥ 64 | 99 [93.5 to 99.97] | 45 [34.8 to 56.4]
  Men W, ≥ 128: number analyzed (Participants) | 83 | 88
  Men W, ≥ 128 | 89 [80.4 to 94.9] | 24 [15.4 to 34.1]
  Men Y, ≥ 8 | 100 [96 to 100] | 61 [50.4 to 71.6]
  Men Y, ≥ 16 | 100 [96 to 100] | 56 [44.7 to 66.3]
  Men Y, ≥ 32 | 95 [87.6 to 98.2] | 44 [33.7 to 55.3]
  Men Y, ≥ 64 | 81 [71.8 to 88.7] | 27 [18.3 to 37.8]
  Men Y, ≥ 128 | 65 [54.1 to 74.6] | 14 [7.2 to 22.6]

21. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against the N. Meningitidis Serogroup A, C, W and Y ≥8, ≥ 16, ≥ 32, ≥ 64, ≥128 at 4 Months After the 3-dose Vaccination Series
Description: The immunogenicity of three doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 against serogroups A, C, W, Y, at 4 months after the 3-dose vaccination series.
Time Frame: At Month 10 (4 months after the 3-dose vaccination series)
Population: Analysis was performed on FAS-Immunogenicity (Month 10)- included all screened subjects who provided consent & demographic &/or baseline screening assessments, received a subject ID & vaccination, & provided evaluable serum samples at Month 10 & whose immunogenicity assay result was available for at least one serogroup A, C, W and Y test strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 86 | 91
Percentage of subjects
  Men A, ≥ 8: number analyzed (Participants) | 85 | 88
  Men A, ≥ 8 | 86 [76.6 to 92.5] | 25 [16.4 to 35.4]
  Men A, ≥ 16: number analyzed (Participants) | 85 | 88
  Men A, ≥ 16 | 84 [73.9 to 90.7] | 23 [14.5 to 32.9]
  Men A, ≥ 32: number analyzed (Participants) | 85 | 88
  Men A, ≥ 32 | 72 [61 to 81] | 18 [10.8 to 27.8]
  Men A, ≥ 64: number analyzed (Participants) | 85 | 88
  Men A, ≥ 64 | 46 [35 to 57] | 8 [3.3 to 15.7]
  Men A, ≥128: number analyzed (Participants) | 85 | 88
  Men A, ≥128 | 14 [7.5 to 23.4] | 7 [2.5 to 14.3]
  Men C, ≥ 8: number analyzed (Participants) | 86 | 89
  Men C, ≥ 8 | 100 [95.8 to 100] | 65 [54.3 to 75]
  Men C, ≥ 16: number analyzed (Participants) | 86 | 89
  Men C, ≥ 16 | 98 [91.9 to 99.72] | 48 [37.6 to 59.2]
  Men C, ≥ 32: number analyzed (Participants) | 86 | 89
  Men C, ≥ 32 | 97 [90.1 to 99.3] | 34 [24 to 44.5]
  Men C, ≥ 64 | 86 [76.9 to 92.6] | 26 [17.1 to 36.2]
  Men C, ≥ 128 | 74 [63.9 to 83.2] | 16 [8.9 to 25]
  Men W, ≥ 8: number analyzed (Participants) | 85 | 83
  Men W, ≥ 8 | 99 [93.6 to 99.97] | 75 [64 to 83.6]
  Men W, ≥ 16: number analyzed (Participants) | 85 | 83
  Men W, ≥ 16 | 98 [91.8 to 99.71] | 66 [55.1 to 76.3]
  Men W, ≥ 32: number analyzed (Participants) | 85 | 83
  Men W, ≥ 32 | 94 [86.8 to 98.1] | 58 [46.5 to 68.6]
  Men W, ≥ 64: number analyzed (Participants) | 85 | 83
  Men W, ≥ 64 | 75 [64.7 to 84] | 36 [25.9 to 47.4]
  Men W, ≥ 128: number analyzed (Participants) | 85 | 83
  Men W, ≥ 128 | 52 [40.7 to 62.7] | 18 [10.5 to 28]
  Men Y, ≥ 8 | 91 [82.5 to 95.9] | 58 [47.4 to 68.5]
  Men Y, ≥ 16 | 86 [76.9 to 92.6] | 51 [39.9 to 61.2]
  Men Y, ≥ 32 | 77 [66.4 to 85.2] | 38 [28.4 to 49.2]
  Men Y, ≥ 64 | 62 [50.5 to 71.9] | 20 [12.2 to 29.4]
  Men Y, ≥ 128 | 40 [29.2 to 50.7] | 9 [3.9 to 16.6]

22. Secondary Outcome: Number of Subjects Reporting Any Solicited Local or Systemic Adverse Events (AEs)
Description: Number of subjects reporting any solicited local or systemic AEs from Day 1 (6 hours) to Day 7 after any meningococcal vaccination is reported. Assessed solicited local symptoms were induration, erythema and pain. Assessed solicited general symptoms were fatigue, myalgia, arthralgia, headache, fever, chills and loss of appetite. Other solicited data included prevention of pain/fever and treatment of pain/fever. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: Day 1 (6 hours) to Day 7 after vaccination
Population: Analysis was performed on Safety Set (solicited AEs & other solicited reactions)-included all screened subjects who provided consent & demographic &/or baseline screening assessments, received a subject ID & a study vaccination, & provided post-vaccination reactogenicity data.
Measure: Count of Participants; unit: Participants
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 90 | 87
Participants
  Any | 62 | 25
  Any Local Reactions | 60 | 15
  Any Systemic Reactions | 27 | 15
  Induration (mm): number analyzed (Participants) | 88 | 87
  Induration (mm) | 6 | 0
  Erythema (mm): number analyzed (Participants) | 87 | 86
  Erythema (mm) | 6 | 0
  Pain: number analyzed (Participants) | 88 | 87
  Pain | 59 | 15
  Nausea: number analyzed (Participants) | 87 | 87
  Nausea | 5 | 5
  Fatigue: number analyzed (Participants) | 87 | 87
  Fatigue | 14 | 11
  Myalgia: number analyzed (Participants) | 87 | 85
  Myalgia | 13 | 3
  Arthralgia: number analyzed (Participants) | 86 | 85
  Arthralgia | 9 | 0
  Headache: number analyzed (Participants) | 88 | 87
  Headache | 13 | 9
  Fever: number analyzed (Participants) | 90 | 85
  Fever | 0 | 1
  Chills: number analyzed (Participants) | 88 | 87
  Chills | 2 | 3
  Loss of appetite: number analyzed (Participants) | 88 | 87
  Loss of appetite | 3 | 3
  Prevention of pain/fever: number analyzed (Participants) | 85 | 84
  Prevention of pain/fever | 0 | 0
  Treatment of pain/fever: number analyzed (Participants) | 85 | 84
  Treatment of pain/fever | 12 | 3

23. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: The number of subjects reporting unsolicited AEs after any vaccination is reported. An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Day 1 to Day 30 after any vaccination
Population: Analysis was performed on Safety set (unsolicited AEs)- included all screened subjects who provided informed consent & demographic and/or baseline screening assessments, received a subject ID and a study vaccination, and had post-vaccination unsolicited adverse event records.
Measure: Count of Participants; unit: Participants
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 93 | 93
Participants | 14 | 11

24. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs), Medically-attended AEs and AEs Leading to Premature Withdrawal.
Description: The number of subjects reporting any SAEs, medically-attended AEs and AEs leading to premature withdrawal during the entire study period is reported. SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any was defined as the occurrence of any unsolicited AE regardless of intensitygrade or relation to vaccination.
Time Frame: During the entire study period (from Day 0 up to Month 10)
Population: Analysis was performed on Safety Set (overall)- included all screened subjects who provide informed consent and demographic and/or baseline screening assessments, received a subject ID and a study vaccination, and have either post-vaccination reactogenicity data or post-vaccination unsolicited adverse event records.
Measure: Count of Participants; unit: Participants
Arm/Group | MenABCWY Group | MenACWY Group
Number analyzed (Participants) | 95 | 94
Participants
  Any SAEs: number analyzed (Participants) | 93 | 93
  Any SAEs | 0 | 0
  Any Medically Attended AEs: number analyzed (Participants) | 93 | 93
  Any Medically Attended AEs | 14 | 20
  Any AEs leading to premature withdrawal | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general AEs were collected from Day 1 to Day 7. Unsolicited AEs were collected from Day 1 to Day 30. SAEs, medically-attended AEs and AEs leading to withdrawal are collected for the entire duration of the study (from Day 0 to Month 10).
Description: Data are presented in terms of number of subjects reporting AEs. The total number of subjects at risk for the frequent adverse events were analysed from the exposed set and the number of subjects at risk for each of the adverse event were analysed from the overall safety set. Therefore, the number of subjects at risk for each adverse event is lesser than the total number of subjects at risk.
Arm/Group | MenABCWY Group | MenACWY Group
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/94
Other Adverse Events (participants affected / at risk) | 63/95 | 27/94
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MenABCWY Group (N=95) | MenACWY Group (N=94)
Headache (Nervous system disorders) | 14/93 (25) | 9/93 (27)
Fatigue (General disorders) | 14/93 (32) | 11/93 (24)
Injection site erythema (General disorders) | 16/93 (44) | 4/93 (12)
Injection site induration (General disorders) | 16/93 (57) | 3/93 (10)
Injection site pain (General disorders) | 60/93 (155) | 15/93 (23)
Nausea (Gastrointestinal disorders) | 5/93 (9) | 5/93 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9/93 (21) | 1/93 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 13/93 (33) | 3/93 (10)
Upper respiratory tract infection (Infections and infestations) | 6/93 (6) | 1/93 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.